CLINICAL TRIAL: NCT05355662
Title: Prognosis Analysis of Elderly Donor Liver From Donation After Cardiac Death in Liver Transplantation: a Multicenter Clinical Study
Brief Title: Prognosis Analysis of Elderly Donor Liver in Liver Transplantation
Status: Completed | Type: Observational
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Principal Investigator, Hu Liangshuo, Principal Investigator, First Affiliated Hospital Xi'an Jiaotong University
Other Study IDs: No. XJTU1AF-CRF-2019-029
Record Dates: First submitted 2022-03-16; First posted 2022-05-02 (Actual); Last update posted 2022-05-02 (Actual); Status verified 2022-03

CONDITIONS: Liver Transplantation; Hepatocellular Carcinoma; Survival
Keywords: elderly donor; liver transplantation; donation after cardiac death; hepatocellular carcinoma; survival
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Aging

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- OLDs: Older liver donors (OLDs) and recipients were defined as individuals whose donor age was equal to or greater than 60 years. Subjects matching the characteristics of this group were screened from the database according to inclusion and exclusion criteria, and preoperative and postoperative characteristics of the corresponding recipients and donors were collected and recorded for subsequent analysis.
  Interventions: Other: Age
- ILDs: Ideal or young liver donors (ILDs) and recipients were defined as donors aged 18-40 years. Subjects matching the characteristics of this group were screened from the database according to inclusion and exclusion criteria, and preoperative and postoperative characteristics of the corresponding recipients and donors were collected and recorded for subsequent analysis.
  Interventions: Other: Age
- ALDs: Average liver donors (ALDs) and recipients were defined as donor age 40-59 years. Subjects matching the characteristics of this group were screened from the database according to inclusion and exclusion criteria, and preoperative and postoperative characteristics of the corresponding recipients and donors were collected and recorded for subsequent analysis.
  Interventions: Other: Age

INTERVENTIONS:
Other: Age — The study was retrospective and did not involve the application of interventions.

SUMMARY:
Based on the follow-up data of elderly donation after cardiac death(DCD) donor liver transplant recipients from the CLTR, a database and official website for national data gathering. patients who met the enrollment criteria were screened for postoperative complications and survival for statistical analysis to understand the prognosis of patients and analyze the risk factors affecting their prognosis.

DETAILED DESCRIPTION:
Since the Chinese organ donation system was developed in 2015, donation has been the only source of organs for transplantation in China. Adult patients (age 18 or older) who underwent LT using grafts from deceased donors between January 1st, 2015, and December 31st, 2018, were retrospectively identified using the CLTR, a database and official website for national data gathering. Based on the follow-up data of elderly DCD donor liver transplant recipients from the CLTR, a database and official website for national data gathering. patients who met the enrollment criteria were screened for postoperative complications and survival for statistical analysis to understand the prognosis of patients and analyze the risk factors affecting their prognosis.

ELIGIBILITY:
Inclusion Criteria:

1. Recipient age ≥ 18 years and < 65 years.
2. Donor age ≥ 18 years.

Exclusion Criteria:

1. Recipient age <18 years or ≥65 years.
2. Donor age <18 years.
3. Patients who died within 30 days after transplantation.
4. Secondary liver transplantation.
5. Multiple organ transplantation.
6. Patients with incomplete data or failed follow-up.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (age 18 or older) who underwent LT using grafts from deceased donors between January 1st, 2015, and December 31st, 2018, were retrospectively identified using the CLTR, a database and official website for national data gathering.
Sampling Method: Non-Probability Sample
Enrollment: 11569 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Post-operative survival time | Time from the end of liver transplantation to the patient's death, or the end of follow-up by December 31, 2020. whichever came first, assessed up to 72 months.
  Postoperative survival time for patients receiving liver transplantation
Transplanted liver status | Time from the end of liver transplantation to the patient's death, or the end of follow-up by December 31, 2020. whichever came first, assessed up to 72 months.The functional status of the transplanted liver was recorded during this period.
  Postoperative Liver Function in Patients Undergoing Liver Transplantation
Recurrence of the primary disease after surgery | The time period between liver transplantation and the initial examination revealing a recurrence of primary disease, or until the end of follow-up on December 31, 2020.whichever came first, assessed up to 72 months.
  Recurrence of primary disease in patients who underwent liver transplantation after surgery

SECONDARY OUTCOMES:
Surgery details | Intraoperative
  Detailed information such as operation time
Post-operative complications in patients who underwent liver transplantation | Time from the end of liver transplantation to the patient's death, or the end of follow-up by December 31, 2020. whichever came first, assessed up to 72 months.During this period, all postoperative complications of the patient will be recorded.
  Specific details of all post-operative complications in patients who underwent liver transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Bo Wang, MD PhD, Study Chair — First Affiliated Hospital Xi'an Jiaotong University

IPD SHARING:
Plan to Share IPD: No
The study was based on national information from the Chinese Liver Transplant Registry and the investigators did not have access to patient information or raw data.